CLINICAL TRIAL: NCT07260851
Title: An Open-label, Randomized, Fasting, Single-dose, 2-sequence, 2-period, Crossover Phase 1 Study to Evaluate the Pharmacokinetics and the Safety After Administration of "DWJ1622" and Co-administration of "DWC202313" and "DWC202314" in Healthy Volunteers
Brief Title: Bioequivalence Study for the Safety and the Pharmacokinetics of DWJ1622, DWC202313, and DWC202314 in Healthy Volunteers Under Fasting Conditions
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DW_DWJ1622102
Record Dates: First submitted 2025-11-16; First posted 2025-12-03 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DWJ1622 (Experimental)
  Interventions: Drug: DWJ1622; Drug: DWC202313, DWC202314
- DWC202313, DWC202314 (Experimental)
  Interventions: Drug: DWJ1622; Drug: DWC202313, DWC202314

INTERVENTIONS:
Drug: DWJ1622 — DWJ1622 (single oral dose) is administered in accordance with the study protocol.
Drug: DWC202313, DWC202314 — DWC202313, DWC202314(single oral dose) is administered in accordance with the study protocol.

SUMMARY:
This study aims to evaluate the safety and pharmacokinetic characteristics of DWJ1622, DWC202313, and DWC202314 in healthy adult volunteers under fasting conditions.

DETAILED DESCRIPTION:
This is an open-label, randomized, oral, single-dose, 2-sequence, 2-period, crossover Phase 1 study designed to compare the pharmacokinetics and safety profiles of DWJ1622 with the co-administration of DWC202313 and DWC202314 in healthy volunteers under fasting conditions. Subjects will be randomized to receive either DWJ1622 or the co-administration of DWC202313 and DWC202314 in different sequences across two study periods with an appropriate washout period.

The primary pharmacokinetic endpoints include the maximum observed plasma concentration (Cmax) and the area under the plasma concentration-time curve to the last measurable concentration (AUClast) of each study drug. Secondary endpoints include the area under the plasma concentration-time curve extrapolated to infinity (AUCinf), the ratio of AUClast to AUCinf (AUClast/AUCinf), the time to reach maximum plasma concentration (Tmax), and the terminal elimination half-life (t1/2). Safety will be evaluated based on adverse events and clinical laboratory tests.

ELIGIBILITY:
Inclusion Criteria:

* Over 19 year old
* Healthy adult volunteers

Exclusion Criteria:

* with a history of mental disorder
* For female volunteers, those who are suspected of being pregnant or lactating

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-11-05 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Cmax | At pre-dose (0 hours), and post-dose 1 to 72 hours.
  Cmax of DWJ1622 and DWC202313, DWC202314
AUClast | At pre-dose (0 hours), and post-dose 1 to 72 hours.
  AUClast of DWJ1622 and DWC202313, DWC202314

SECONDARY OUTCOMES:
AUCinf | At pre-dose (0 hours), and post-dose 1 to 72 hours.
  AUCinf of DWJ1622 and DWC202313, DWC202314
AUClast/AUCinf | At pre-dose (0 hours), and post-dose 1 to 72 hours.
  AUClast/AUCinf of DWJ1622 and DWC202313, DWC202314

CONTACTS AND LOCATIONS:
Locations (1):
- H Plus YANGJI Hospital, Seoul, Gwanak-gu, South Korea